CLINICAL TRIAL: NCT03499457
Title: Penicillin Allergy in Shfayim Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Dr. Lital Goldberg, dr lital goldberg, Clalit Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0185-17-COM2
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Penicillin Allergy
Keywords: Penicillin Allergy; chalenge test; primary clinic
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): penicillin chalange test, as descibed.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — chalange test of 50 mg, and after an hour 500 mg

SUMMARY:
revising penicillin allergy in the medical records, by taking full medical history and giving a challange test, in order to imrove the medical records and treatment possibilities.

DETAILED DESCRIPTION:
issuing a list of patients with a title of penicillin allergy in their medical record. inviting these patients to an appointmnet with their family physician, in which a specific history will be take to evaluate the quality of the allergy.

patients with suscpition of a life threatening allergic reaction will be reffered to an allergy clinic for the challange test. the rest of the pateints will be given the test in the primary clinic: 1ml (50 grams) of amoxicillin, and an hour later a full dose of 500 mg amoxicillin.

after determining no allergic reaction develops the title will be erased from the medical record.

ELIGIBILITY:
Inclusion Criteria:

penicillin allergy in the medical record

Exclusion Criteria:

pregnancy lack of informed consent

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
immidiate urticarial reaction | with 2 hours of test
  shortness of breath, angioedema

SECONDARY OUTCOMES:
rash | with 2 hours of test
  body rash or itch seen by patient or physician

CONTACTS AND LOCATIONS:
Overall Officials: lital f goldberg, MD. MPH, Principal Investigator — Clalit Health Services